CLINICAL TRIAL: NCT04677452
Title: An Open-Label Phase 1 Dose Exploration Study of JWCAR129, BCMA-targeted Chimeric Antigen Receptor (CAR) T Cells, in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Dose Exploration Study OF JWCAR129, BCMA-Targeted CART for RRMM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR129
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Safety and Efficacy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR129 (Experimental): Subjects will receive a course of lymphodepleting chemotherapy with fludarabine and cyclophosphamide followed by a single dose of JWCAR129
  Interventions: Biological: JWCAR129

INTERVENTIONS:
Biological: JWCAR129 — Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JWCAR129. During JWCAR129 production, participants may receive bridging chemotherapy for disease control. Following successful generation of JWCAR129 product, participants will receive a course of lymphodepleting chemotherapy followed by one dose of JWCAR129 administered intravenously (IV).

SUMMARY:
This is an open-label, Phase 1 dose exploration study to evaluate the safety and tolerability and to determine recommended Phase 2 dose(s) of JWCAR129, a CAR T-cell product that targets B-cell maturation antigen (BCMA), in adult subjects with relapsed and/or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above.
2. Signed the Informed Consent Form.
3. Diagnosis of multiple myeloma (MM) with relapsed and/or refractory disease. Subjects must have received at least 3 prior anti-myeloma treatment regimens (note: induction with or without bone marrow transplant and with or without maintenance therapy is considered one regimen). Subjects must be refractory to the last anti-myeloma treatment regimen prior to entering the study.

   1. Autologous hematopoietic stem cell transplantation.
   2. A regimen that included an immunomodulatory agent (eg, thalidomide, lenalidomide, pomalidomide) and a proteasome inhibitor (eg, bortezomib, carfilzomib, ixazomib), either alone or in combination. Subjects must have undergone at least 2 consecutive cycles of treatment for each regimen unless progressive disease was the best response to the regimen.
   3. Anti-CD38 (eg, daratumumab) as part of a combination regimen or as a monotherapy.

   Subjects who were not candidates to receive one or more of the above treatments (ie, contraindicated) are eligible; the reason for not receiving treatment must be clearly documented in the case report form.
4. Subjects must have measurable disease.
5. Subject must be willing to provide fresh bone marrow biopsy samples during Screening (and prior to study treatment, if required).
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Adequate renal, bone marrow, hepatic, pulmonary, and cardiac function

Exclusion Criteria:

1. Subjects with known active or history of CNS involvement by malignancy
2. Subjects with solitary plasmacytoma; active or history of plasma cell leukemia (PCL); Waldenstrom's macroglobulinemia; Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal plasmaproliferative disorder, Skin changes (POEMS) syndrome; or symptomatic amyloidosis
3. History of another primary malignancy that has not been in remission for at least 3 years. The following are exempt from the 3-year limit: non-melanoma skin cancer, curatively treated localized prostate cancer, cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Pap smear, and in situ breast cancer that has been completely resected.
4. Require systemic immunosuppressive therapies (eg, calcineurin inhibitors, methotrexate, mycophenolate, rapamycin, thalidomide, immunosuppressive antibodies such as anti-IL-6 or anti-IL-6 receptor [IL-6R])
5. Prior CAR T-cell or other genetically-modified T-cell therapy
6. Prior treatment with a BCMA-targeted agent
7. History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
8. Untreated or active infection at time of initial screening, at the time of leukapheresis, within 72 hrs before lymphodepletion, or 5 days before JWCAR129 infusion.
9. History of any of the following cardiovascular conditions within 6 months of initial screening: Class III or IV heart failure as defined by the New York Heart Association (NYHA), myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant cardiac disease
10. History of severe immediate hypersensitivity reaction to any of the protocol-mandated or recommended agents used in this study
11. Allogeneic hematopoietic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | 28 days
  Proportion of subjects with adverse events meeting DLT criteria
Incidence and severity of adverse events | 2 years
  Proportion of subjects with adverse events overall and by severity grade
Incidence and severity of clinically significant laboratory abnormalities | 2 years
  Proportion of subjects with clinically significant laboratory abnormalities overall and by severity grade

SECONDARY OUTCOMES:
Cmax | 2 years
  Maximum concentration (Cmax) of JWCAR129 in the blood
Tmax | 2 years
  Time to maximum concentration (Tmax) of JWCAR129 in the blood
AUC | 2 years
  Area under the concentration vs time curve (AUC) of JWCAR129 in the blood
Duration of persistence | 2 years
  Duration of persistence of JWCAR129 CAR T cells in the blood
Overall response rate | 2 years
  Proportion of subjects with a partial response (PR) or better by IMWG criteria
CR rate | 2 years
  Proportion of subjects with a CR by IMWG criteria

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China